CLINICAL TRIAL: NCT00137878
Title: A Phase II Randomized Trial Comparing TNFerade™ Biologic With Capecitabine and Radiation Therapy Followed by Surgical Resection Versus Capecitabine and Radiation Therapy Followed by Surgical Resection for the Treatment of Rectal Cancer
Brief Title: TNFerade™ Plus Chemo/Radiation/Surgery for Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GenVec (Industry)
Responsible Party: Paul Fischer, PhD, GenVec
Allocation: Randomized | Purpose: Treatment
Other Study IDs: GV-001.007; NCT00069147 (obsolete NCT alias); NCT00072241 (obsolete NCT alias)
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2011-05

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

INTERVENTIONS:
Drug: TNFerade™

SUMMARY:
The purpose of this study is to determine if the addition of TNFerade™ to pre-operative chemoradiotherapy increases the number of pathologic complete responses when compared to pre-operative chemoradiotherapy alone as assessed following complete surgical resection of primary rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have biopsy proven T3 or T4 rectal cancer which is confined to the primary tumor site with or without regional lymph node involvement
* Patients must be willing to return for follow-up
* Patients must be able to give and sign informed consent
* Patients must be suitable candidates for surgical resection post-chemoradiation, i.e. no history of severe congestive heart failure or severe pulmonary disease
* Life expectancy > 6 months

Exclusion Criteria:

* Patients with evidence of distant metastatic disease
* Any of the following hematologic abnormalities: hemoglobin (HGB) < 8.0 gm/dL unable to be corrected with a transfusion; absolute neutrophil count (ANC) < 1500 cells/mm3; platelets < 100,000/mm3; activated partial thromboplastin time (APTT) ratio or International Normalized Ratio (INR) > 1.5 (except in patients who are therapeutically anticoagulated for non-related medical conditions such as atrial fibrillation and whose anti-thrombotic treatment cannot be withheld for vector injection or surgery).
* A history of hepatic cirrhosis or present hepatic dysfunction with total bilirubin > 2.0 mg/dL except for patients with Gilbert's syndrome who must have a direct bilirubin </= 1.0 mg/dL; AST/ALT >/= 2.5 times upper limit of normal.
* Renal insufficiency as determined by a serum creatinine > 2.0 mg/dL
* Patients may not have received prior therapy with chemotherapy, biologic therapy or radiation therapy for rectal cancer
* Significant history of a medical problem that would preclude the patient from undergoing an operative procedure such as a history of severe congestive heart failure or active ischemic heart disease
* Concurrent second malignancy requiring systemic therapy
* Pregnant or lactating women
* Chronic systemic corticosteroid use
* Prior surgery for rectal cancer
* Patients with history of deep venous thrombosis or pulmonary embolism
* Patients with Doppler evidence of deep venous thrombosis at screening
* Known history of documented coagulopathy or thrombophilic disorders
* Hormone replacement therapy within one month prior to Day 1
* Known history of documented cerebrovascular disease, stroke or transient ischemic attack (TIA)
* Surgery within the last one month, excluding diverting colostomy or ileostomy for obstruction

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Cancer Research, NCI, Bethesda, Maryland, United States

REFERENCES:
- See also: PubMed.gov — http://www.ncbi.nlm.nih.gov/pubmed?term=A%20Pilot%20Feasbility%20Study%20of%20TNFerade%20Biologic%20with%20Capecitabine%20and%20Radiation%20Therapy